CLINICAL TRIAL: NCT03253809
Title: Survey of QRS Frequency at Various Left Ventricular Pacing Sites for Cardiac Resynchronization
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Issue with trial administration/conduct
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17-650
Record Dates: First submitted 2017-08-16; First posted 2017-08-18 (Actual); Results first posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Cardiomyopathies; Congestive Heart Failure
MeSH Terms: conditions — Cardiomyopathies; Heart Failure

STUDY DESIGN:
Intervention Model Description: Nonrandomized survey of different pacing sites in the coronary veins.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Coronary Sinus Branch Pacing (Experimental): After cannulation, pacing impulses will be delivered via a Biotronik Vision Guidewire to 3 sites (apical, mid ventricular, and basal) within each coronary sinus branch receiving venous blood from the anterior, lateral and posterior regions of the ventricle.
  ECG signals will be saved digitally for analysis
  Interventions: Device: Biotronik Vision Guidewire

INTERVENTIONS:
Device: Biotronik Vision Guidewire — The apical, mid ventricular and basal sites within the anterior,posterior and lateral coronary sinus branch veins will be paced.

SUMMARY:
LV pacing at various sites with recording of ECG and subsequent signal analysis at different sites.

DETAILED DESCRIPTION:
During routine cardiac resynchronization pacemaker or implantable defibrillator (ICD) implantation (including de-novo and upgrade from standard device, additional pacing within 3 different coronary veins will be performed in combination with a previously implanted right ventricular pacing or ICD lead. The resulting electrocardiogram signal will be analyzed afterwards. A time-frequency analysis (TFA) of several ECG leads at each paced site will be performed and compared. The results of the TFA analysis will not be used to select pacing lead location in this study.

The patient will then receive the left ventricular pacing lead in the standard manner.

ELIGIBILITY:
Inclusion Criteria:

* Standard implantation for cardiac resynchronization ICD or PM implantation
* Cardiomyopathy with LVEF <35%
* QRS duration greater than 120 msec

Exclusion Criteria:

- Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Niebauer, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Coronary Sinus Branch Pacing: After cannulation, pacing impulses will be delivered via a Biotronik Vision Guidewire to 3 sites (apical, mid ventricular, and basal) within each coronary sinus branch receiving venous blood from the anterior, lateral and posterior regions of the ventricle.
  ECG signals will be saved digitally for analysis
  Biotronik Vision Guidewire: The apical, mid ventricular and basal sites within the anterior,posterior and lateral coronary sinus branch veins will be paced.
Period: Overall Study
Arm/Group | Coronary Sinus Branch Pacing
Started | 14
Completed | 0
Not Completed | 14
Not completed — Unable to obtain study related data | 14

BASELINE CHARACTERISTICS:
Arm/Group | Coronary Sinus Branch Pacing
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 13
  African American | 1
Need for implantation of a left ventricular pacing lead via the coronary sinus branch beins [Count of Participants; unit: Participants] | 14

OUTCOME MEASURES:

1. Primary Outcome: QRS Frequency at Each Paced Location
Description: Time frequency analysis performed at each location
Time Frame: Baseline
Population: Unable to collect or analyze the data. Study was not feasible.
Arm/Group | Coronary Sinus Branch Pacing
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Day of the index procedure
Arm/Group | Coronary Sinus Branch Pacing
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-05-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT03253809/Prot_000.pdf
  • Informed Consent Form (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT03253809/ICF_001.pdf